CLINICAL TRIAL: NCT01634451
Title: Development and Evaluation of Strategies to Improve Sedation Quality in InTensive Care
Acronym: DESIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2012/R/AN/01
Record Dates: First submitted 2012-06-20; First posted 2012-07-06 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Critical Illness
Keywords: Sedation; Quality
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Education Package (Active Comparator): 2 ICUs; one large and one small. Randomised to receive bespoke education package for the 9 month intervention period
  Interventions: Other: Bespoke on-line sedation education package
- Education and Feedback (Active Comparator): 2 ICUs; one large and one small. Randomised to receive a bespoke education package and real-time,site specific, outcome process feedback they will disseminate to their staff for the 9 month intervention period.
  Interventions: Other: Sedation specific outcome process feedback
- Education and Sedation Monitoring (Active Comparator): 2 ICUs; one large and one small. Randomised to receive a bespoke education package and a new novel sedation (responsiveness) monitor for the 9 month intervention period.
  Interventions: Device: Responsiveness monitoring; novel sedation monitor
- Education, Feedback, Sedation Monitoring (Active Comparator): 2 ICUs; one large and one small. Randomised to receive a bespoke education package, real-time,site specific, outcome process feedback they will disseminate to their staff and a new novel sedation (responsiveness) monitor for the 9 month intervention period.
  Interventions: Other: Sedation specific outcome process feedback; Device: Responsiveness monitoring; novel sedation monitor

INTERVENTIONS:
Other: Bespoke on-line sedation education package — A bespoke on-line education package has been developed and will be accessible by all ICU nursing staff. They will have unique logins and the system will track their use and completion of the education package. There is a small multiple choice assessment at the end of the package.
  Other Names: Bespoke Education Package
  Arms: Education Package
Other: Sedation specific outcome process feedback — Using statistical process charts, the data gathered from the Sedation quality Tools (SQATs) completed each shift by the ICU nurses, will be fed back highlighting sedation specific outcomes e.g. number of over sedated days per 1000 ventilator days.
  Other Names: Sedation pecific outcome process feedback
  Arms: Education and Feedback; Education, Feedback, Sedation Monitoring
Device: Responsiveness monitoring; novel sedation monitor — Responsiveness monitoring (developed by GE Healthcare) is a novel technology used to monitor patient responsiveness and essentially alert ICU nursing staff when their patients may be over sedated.
  Other Names: Responsiveness Monitoring
  Arms: Education and Sedation Monitoring; Education, Feedback, Sedation Monitoring

SUMMARY:
Intensive Care Units (ICUs) across Scotland are working with the Scottish Patient Safety Programme (SPSP) to reduce healthcare associated infections (HAls). This is being done through implementation of "care bundles". Ensuring that ICU patients get the correct amount of sedation (medicine that makes patients sleepy) is part of this bundle, but is proving the most difficult to get right. It's important healthcare staff (nurses and doctors) get sedation levels correct because too much sedation is linked with increased hospital acquired infections (HAIs), longer intensive care (ICU) and hospital stays, and possibly higher death rates. This quality improvement project will develop and introduce three interventions that may improve sedation practice: first, an ICU sedation education package; second, feedback of sedation-related performance data (graphs and charts); and third, introduction of a CE (Conformité Européenne - With the CE marking on a product, the manufacturer ensures that the product conforms with the essential requirements of European regulations) marked new technology designed to improve sedation management. The investigators will study the effect these interventions, in different combinations, have on sedation management and quality in the participating ICUs. Eight ICUs in Scotland will take part in the project, pairs (2 ICUs) will be assigned randomly to different combinations as follows: 1.Enhanced education alone, 2. Education plus process/outcome measure feedback (graphs and charts), 3. Education plus introduction of a new sedation monitoring technology, or 4. Education,process/outcome measure feedback, and sedation monitoring technology. The investigators will evaluate which combinations of education, feedback, and technology provide the most patient benefit in the NHS. In addition both nursing & medical staff will be observed in clinical practice & interviewed about their clinical practice to increase understanding about sedation management from different view points and inform the education package content. These data will also help implement the findings after the research is completed if a benefit is found.

ELIGIBILITY:
Inclusion Criteria:

1. All patients admitted to ICU mechanically ventilated and intubated.
2. All patients in whom mechanical ventilation via an endotracheal tube is instituted at some time after ICU admission will also be eligible for inclusion from the time intubation and mechanical ventilation begins.

Exclusion Criteria:

1. Patients who are not receiving mechanical ventilation via an endotracheal tube
2. Patients who received mechanical ventilation following ICU admission but this has been discontinued at the time of screening for study inclusion
3. Patients in whom discontinuation of mechanical ventilation is anticipated in the next 4 hours
4. Patients in whom a decision to withdraw active therapy has been made
5. Patients who have already been enrolled in the during the same hospital admission
6. Patients whom have been mechanically ventilated and intubated for greater than 24 hrs by the time relatives are approached for consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1637 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline the effect of individual and combinations of the interventions named on achievement of optimal sedation practice | Cluster trial examining group effects over a 20 month period. Data available June 2014.
  The % of ventilated patient days with optimal sedation will be compared across and between the groups. A sedation quality assessment tool has been developed for the purpose of the study:
  Group 1 -Education package only (bespoke sedation education) Group 2 -Education package and real time (site specific) process feedback about sedation practices Group 3 - Education and responsiveness (sedation) technology Group 4 - Education package, real time (site specific) process feedback about sedation practices and responsiveness (sedation) technology

SECONDARY OUTCOMES:
Number of ventilation days | Cluster trial examining group effects over a 20 month period. Data available June 2014.
ICU stay duration | Cluster trial examining group effects over a 20 month period. Data available June 2014.
Number of days on sedation | Cluster trial examining group effects over a 20 month period. Data available June 2014.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Walsh, MD, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary Edinburgh, Glasgow Royal Infirmary, Monklands Hospital, Victoria Infirmary Glasgow, Forth Valley Royal, Ninewells hospital, Dumfries Infirmary , Victoria Hospital Kirkcaldy, Edinburgh, Glasgow, Airdrie, Larbert, Dumfries, Dundee, United Kingdom

REFERENCES:
- [Derived] Kydonaki K, Hanley J, Huby G, Antonelli J, Walsh TS; Development and Evaluation of Strategies to Improve Sedation practice in inTensive care (DESIST) study investigators. Challenges and barriers to optimising sedation in intensive care: a qualitative study in eight Scottish intensive care units. BMJ Open. 2019 May 24;9(5):e024549. doi: 10.1136/bmjopen-2018-024549. PMID 31129576
- [Derived] Walsh TS, Kydonaki K, Antonelli J, Stephen J, Lee RJ, Everingham K, Hanley J, Phillips EC, Uutela K, Peltola P, Cole S, Quasim T, Ruddy J, McDougall M, Davidson A, Rutherford J, Richards J, Weir CJ; Development and Evaluation of Strategies to Improve Sedation Practice in Intensive Care (DESIST) study investigators. Staff education, regular sedation and analgesia quality feedback, and a sedation monitoring technology for improving sedation and analgesia quality for critically ill, mechanically ventilated patients: a cluster randomised trial. Lancet Respir Med. 2016 Oct;4(10):807-817. doi: 10.1016/S2213-2600(16)30178-3. Epub 2016 Jul 26. PMID 27473760
- [Derived] Walsh TS, Kydonaki K, Antonelli J, Stephen J, Lee RJ, Everingham K, Hanley J, Uutelo K, Peltola P, Weir CJ; Development and Evaluation of Strategies to Improve Sedation practice in in Tensive care Study Investigators. Rationale, design and methodology of a trial evaluating three strategies designed to improve sedation quality in intensive care units (DESIST study). BMJ Open. 2016 Mar 4;6(3):e010148. doi: 10.1136/bmjopen-2015-010148. PMID 26944693